CLINICAL TRIAL: NCT06702943
Title: Comparative Study of the Efficacy and Safety of Tigecycline Based Regimen Versus Colistimethate Sodium-based Regimen in Patients with Central Nervous System Bacterial Infections
Brief Title: Comparing Tigecycline Vs. Colistimethate in CNS Infections
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: ACUC-FP-ASU#265
Record Dates: First submitted 2024-09-10; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-06

CONDITIONS: Central Nervous System Infections
Keywords: Central nervous system infections; MDR bacteria
MeSH Terms: conditions — Central Nervous System Infections | interventions — Tigecycline; colistinmethanesulfonic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Pediatrics patients having EVD and suffering from meningitis caused by MDR bacteria
  Interventions: Drug: Tigecycline (Tygacil); Drug: Colistimethate sodium (CMS)

INTERVENTIONS:
Drug: Tigecycline (Tygacil) — tigecycline-based regimen administered both intravenously (IV) and intraventricularly (IVT) for 14-21 days
Drug: Colistimethate sodium (CMS) — Colistimethate sodium-based regimen (standard therapy for MDR infections) administered both IV and IVT for 14-21 days.

SUMMARY:
This observational study compares the efficacy and safety of tigecycline, an alternative antibiotic with broad-spectrum activity, versus the standard colistimethate sodium-based regimen in managing these infections in pediatric patients.

Inclusion Criteria:

Pediatric patients aged 1 month to 18 years. Presence of CNS infection symptoms such as fever, altered mental status, and positive cerebrospinal fluid (CSF) findings.

EVD placement for managing CNS infections.

Exclusion Criteria:

Known allergy to tigecycline or colistimethate sodium. Patients with concurrent severe comorbid conditions that may confound study results.

Neonates (less than 1 month old), pregnant, or breastfeeding patients.

Outcome Measures:

Primary Outcomes: Clinical cure (resolution of infection symptoms) and microbiological cure (sterilization of CSF cultures).

Secondary Outcomes: Mortality rates and adverse drug events, such as nephrotoxicity, hepatotoxicity, chemical meningitis, or seizures.

DETAILED DESCRIPTION:
Background:

Central nervous system (CNS) bacterial infections, such as meningitis and ventriculitis, are severe conditions in pediatric patients, often resulting from healthcare-associated complications, invasive procedures, or the spread of infection from other body sites. Multi-drug-resistant (MDR) pathogens, particularly carbapenem-resistant Acinetobacter baumannii, pose significant challenges in treating these infections. Standard treatment options, like colistimethate sodium, are associated with limited penetration into the CNS and potential toxicity. This study compares the efficacy and safety of tigecycline, an alternative antibiotic with broad-spectrum activity, versus the standard colistimethate sodium-based regimen in managing these infections in pediatric patients.

Data Collection and Analysis:

Patient data, including demographics, clinical presentations, treatment regimens, laboratory findings (CSF analysis, cultures), and adverse effects, will be systematically collected and analyzed. The study will employ appropriate statistical tests to determine the significance of differences between the two groups.

Ethical Considerations:

Ethical approval will be obtained from the Research Ethics Committees of Ain Shams University and Cairo University. Informed consent will be obtained from the guardians of all pediatric patients. The study will ensure strict adherence to ethical guidelines, including patient confidentiality and data protection.

Expected Impact:

This study aims to provide crucial data on the effectiveness and safety of alternative antibiotic regimens for pediatric CNS infections, potentially guiding clinical practice and improving outcomes for children affected by these severe infections in Egypt and globally.

Study Design:

A prospective observational clinical trial conducted on Pediatrics at Cairo University Hospitals, Egypt.

Study Population:

A total of 70 pediatric patients, aged 1 month to 18 years, admitted with confirmed or suspected CNS infections and with an external ventricular drain (EVD) in place.

Patient Groups:

Intervention Group (n = 35): Pediatric patients receiving a tigecycline-based regimen administered both intravenously (IV) and intraventricularly (IVT) for 14-21 days.

Control Group (n = 35): Pediatric patients receiving a colistimethate sodium-based regimen (standard therapy for MDR infections) administered both IV and IVT for 14-21 days.

Data Collection and Analysis:

Patient data, including demographics, clinical presentations, treatment regimens, laboratory findings (CSF analysis, cultures), and adverse effects, will be systematically collected and analyzed. The study will employ appropriate statistical tests to determine the significance of differences between the two groups.

Ethical Considerations:

Ethical approval will be obtained from the Research Ethics Committees of Ain Shams University and Cairo University. Informed consent will be obtained from the guardians of all pediatric patients. The study will ensure strict adherence to ethical guidelines, including patient confidentiality and data protection.

Expected Impact:

This study aims to provide crucial data on the effectiveness and safety of alternative antibiotic regimens for pediatric CNS infections, potentially guiding clinical practice and improving outcomes for children affected by these severe infections in Egypt and globally.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1 month to 18 years.
* Presence of CNS infection symptoms such as fever, altered mental status, and positive cerebrospinal fluid (CSF) findings.
* EVD placement for managing CNS infections.

Exclusion Criteria:

* Known allergy to tigecycline or colistimethate sodium. Patients with concurrent severe comorbid conditions that may confound study results.

Neonates (less than 1 month old).

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 70 pediatric patients, aged 1 month to 18 years, admitted with confirmed or suspected CNS infections and with an external ventricular drain (EVD) in place.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Microbiological eradication | follow up of the patients from time of enrollment to end of treatment is for 14-21 days
  CSF Culture: Conducted at diagnosis and follow up for it till the end of the treatment course to monitor microbiological clearance. Two consecutive negative cultures are required to consider positive microbiological eradication.
Clinical Cure rate | follow up of the patients from time of enrollment to end of treatment is for 14-21 days
  Resolution of infection symptoms like fever, seizures, fatigue and neck stiffness.

IPD SHARING:
Plan to Share IPD: No